CLINICAL TRIAL: NCT04350320
Title: Administration of Colchicine Plus Standard Treatment vs. Standard Therapy, in Hospitalized Patients With COVID-19, Within the First 48 Hours, and no Severity Criteria.
Brief Title: Trial to Study the Benefit of Colchicine in Patients With COVID-19
Acronym: COL-COVID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundacion para la Formacion e Investigacion Sanitarias de la Region de Murcia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMIB-COLVID-2020-03
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: COVID19
MeSH Terms: conditions — COVID-19 | interventions — Colchicine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase III, prospective, randomized, controlled, open-label and pragmatic trial, comparing the administration of colchicine plus standard treatment vs. standard therapy, in hospitalized patients with COVID-19, within the first 48 hours, and no severity criteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- COLCHICINE (Experimental): The colchicine treatment includes an initial dose of 1.5 mg (1 mg and 0.5 mg two hours after), followed by 0.5 mg every 12 hours during the next 7 days and 0.5 mg every 24 hours until the completion of 28 days of total treatment. In patients receiving ritonavir or lopinavir or with reduced renal clearance (<50 ml/min/1.37m2), weight <70 kg or age >75 years old, the dose will be adjusted to the half.
  + standard therapy for COVID-19 according to the stablished hospital protocols.
  Interventions: Drug: Colchicine Tablets; Drug: Standard therapy for COVID-19 according to the stablished hospital protocols.
- control group (Placebo Comparator): Standard therapy for COVID-19 according to the stablished hospital protocols.
  Interventions: Drug: Standard therapy for COVID-19 according to the stablished hospital protocols.

INTERVENTIONS:
Drug: Colchicine Tablets — standard therapy for COVID-19 according to the stablished hospital protocols.
  Arms: COLCHICINE
Drug: Standard therapy for COVID-19 according to the stablished hospital protocols. — standard therapy for COVID-19 according to the stablished hospital protocols.

SUMMARY:
COVID-19 is associated with a cytokine storm that leads to respiratory distress, multiorgan failure and elevated mortality. Oral colchicine exhibits high anti-inflammatory capacity attributed to the inhibition of microtubules polymerization, inflammasome and production of IL-1β and IL-6, which could prevent the inflammatory storm in COVID-19 patients at risk. We present a randomized clinical trial, controlled, open-label and pragmatic, including COVID-19 patients requiring hospitalization but no intensive care yet. Colchicine will be started within the first 48 hours and then administered for four weeks using a descending dose. The benefit will be study in terms of clinical evolution (WHO 7-point scale) and IL-6 levels, as well as other clinical and biochemical secondary end-points. In the case of positive results, the clinical impact would be relevant given that this oral medication is widely accessible which would help to prevent the inflammatory complications associated with COVID-19.

DETAILED DESCRIPTION:
This is a Phase III, prospective, pragmatic, randomized, controlled and open-label trial, comparing standard of care vs. standard of care plus COLCHICINE for four weeks, in patients hospitalized due to COVID-19 and confirmed infection by SARSCov2, within the first 48 hours after the hospital admission. Patients meeting severity criteria will be excluded, defined as established limitation of therapeutic effort or need for invasive mechanical ventilation at the time of inclusion. The colchicine treatment includes an initial dose of 1.5 mg (1 mg and 0.5 mg two hours after), followed by 0.5 mg every 12 hours during the next 7 days and 0.5 mg every 24 hours until the completion of 28 days of total treatment. In patients receiving ritonavir or lopinavir or with reduced renal clearance (<50 ml/min/1.37m2), weight <70 kg or age >75 years old, the dose will be adjusted to the half.

Patients meeting all the inclusion criteria and none of the exclusion ones (see below), after signing the informed consent, will be centrally randomized to "colchicine" or "control" group. Patients in both groups will receive the standard therapy for COVID-19 according to the stablished hospital protocols. Randomization will be controlled by: age, sex, time from initiation of symptoms, cardiovascular disease, the 7 point WHO and levels of C-reactive protein, ferritin, D-dimer, IL-6 and lymphocyte levels.

ELIGIBILITY:
Inclusion Criteria:

1. SARS-CoV-2 infection confirmed by PCR.
2. Admitted in the hospital in the previous 48 hours, with clinical status 3, 4 or 5 of WHO classification.
3. Age above 18 years old.
4. Informed written consent.

Exclusion Criteria:

1. Invasive mechanical ventilation needed.
2. Established limitation of the therapeutic effort
3. Inflammatory bowel disease (IBD: Chron Syndrome or Ulcerative colitis), chronic diarrhea or malabsorption.
4. Previous neuromuscular disease.
5. Other disease with an estimated vital prognosis under 1 year.
6. Severe renal insufficiency (glomerular filtration rate <30 mL/min/1.73m2)
7. Medical records of cirrhosis, active chronic hepatitis or severe hepatic disease defined by GOT or GPT levels three times above the normal upper limit.
8. Patients with previous colchicine treatment for other diseases (mainly chronic prescriptions for familial Mediterranean fever or gout). Clearance period will not be required for patients treated with colchicine who stopped the treatment before the randomization.
9. Patients with history of allergic reaction or significant sensitivity to colchicine.
10. Treatment with immunosuppressive agents, corticoids or interleukine-1 antagonists for 6 months before inclusion.
11. Pregnant or breastfeeding female, confirmed by a positive result in the human chorionic gonadotropin (hCG) test.
12. Fertile woman, or post-menopausal during less than one year and non-surgically sterilized. Women of fertile age may be included if using at least one contraceptive method and preferably two complementary contraceptive methods.
13. Use of other investigational drugs in the moment of inclusion, or during 30 days previous to inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Changes in the patients' clinical status through the 7 points ordinal scale WHO R&D Blueprint expert group | 7,14,28 Days
  improve in the clinical evolution of patients hospitalized
Changes in IL-6 concentrations | up to day 28.
  improve in the clinical evolution of patients hospitalized

SECONDARY OUTCOMES:
Improvement in the clinical status | up to day 28.
  time needed to reduce at least 2 points in the 7-point Ordinal Scale for Clinical Improvement by WHO R&D Blueprint expert group (0-7)
Changes in the score for the Sequential Organ Failure Assessment (SOFA score) | up to day 28.
  Sequential Organ Failure Assessment (SOFA score) (0-14)
Changes in the punctuation in the National Early Warning Score | up to day 28.
  National Early Warning Score (NEWS scale
Number of days with invasive mechanical ventilation | up to day 28.
Number of days with high flow oxygen therapy | up to day 28.
Changes in other inflammatory markers | up to day 28
  C-reactive protein,
Changes in other inflammatory markers | up to day 28
  TNF-alfa,
Changes in other inflammatory markers | up to day 28
  GDF-15,
Changes in other inflammatory markers | up to day 28
  IL-1β
Changes in severity markers | up to day 28
  D-dimer
Changes in severity markers | up to day 28
  leucocytes
Changes in severity markers | up to day 28
  lymphocytes
Changes in severity markers | up to day 28
  platelets
Changes in severity markers | up to day 28
  LDH
Changes in severity markers | up to day 28
  ferritin
Changes in myocardial damage | up to day 28
  myocardial stress markers hsTnT
Changes in myocardial damage | up to day 28
  myocardial stress markers NT-proBNP
Time until reaching a virus negative status | up to day 28
  RT-PCR assay
Length of hospital stay | up to day 28
  Length of hospital stay
Number of days in the intensive care unit. | up to day 28
  Number of days in the intensive care unit.
Mortality | up to day 28
  Mortality

CONTACTS AND LOCATIONS:
Overall Officials: Domingo A Pascual Figal, MD, Principal Investigator — HCUVA
Locations (1):
- Virgen de la Arrixaca University Clinical Hospital, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mikolajewska A, Fischer AL, Piechotta V, Mueller A, Metzendorf MI, Becker M, Dorando E, Pacheco RL, Martimbianco ALC, Riera R, Skoetz N, Stegemann M. Colchicine for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Oct 18;10(10):CD015045. doi: 10.1002/14651858.CD015045. PMID 34658014
- [Derived] Pascual-Figal DA, Roura-Piloto AE, Moral-Escudero E, Bernal E, Albendin-Iglesias H, Perez-Martinez MT, Noguera-Velasco JA, Cebreiros-Lopez I, Hernandez-Vicente A, Vazquez-Andres D, Sanchez-Perez C, Khan A, Sanchez-Cabo F, Garcia-Vazquez E; COL-COVID Investigators. Colchicine in Recently Hospitalized Patients with COVID-19: A Randomized Controlled Trial (COL-COVID). Int J Gen Med. 2021 Sep 11;14:5517-5526. doi: 10.2147/IJGM.S329810. eCollection 2021. PMID 34539185